CLINICAL TRIAL: NCT03374267
Title: Clinical Research Platform On Urologic Cancer Treatment And Outcome (Registry Platform Urologic Cancer; CARAT)
Brief Title: Registry Platform Urologic Cancer
Acronym: CARAT
Status: Recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: iOM-110363
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Renal Cell Carcinoma; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- aRCC: Patients with advanced renal cell carcinoma
  Interventions: Other: Routine care as per site standard.
- aUBC: Patients with advanced urothelial carcinoma (locally advanced and inoperable, or metastatic)
  Interventions: Other: Routine care as per site standard.
- High-risk MIUC: Patients with muscle-invasive urothelial carcinoma classified as high-risk after radical surgery (ypT2-ypT4 and/or ypN+,M0 for patients with prior neoadjuvant chemotherapy; pT3-pT4 and/or pN+, M0 for patients without prior neoadjuvant chemotherapy)
  Interventions: Other: Routine care as per site standard.

INTERVENTIONS:
Other: Routine care as per site standard. — Physician's choice according to patient's needs.

SUMMARY:
The purpose of the project is to set up a national, prospective, longitudinal, multicenter cohort study with associated satellites, a tumor registry platform, to document uniform data on characteristics, molecular diagnostics, treatment and course of disease, to collect patient-reported outcomes and to establish a decentralized biobank for patients with advanced renal cell carcinoma or urothelial cancer in Germany.

DETAILED DESCRIPTION:
CARAT is a national, observational, prospective, longitudinal, multicenter cohort study (tumor registry platform) with the purpose to record information on the antineoplastic treatment of renal cell carcinoma and urothelial cancer in Germany. The registry will follow patients with advanced renal carcinoma for up to three years, and patients with advanced urothelial cancer for up to two years. It will identify common therapeutic sequences and changes in the treatment of the disease. At inclusion, data in patient characteristics, comorbidities, tumor characteristics and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented. Moreover, data on perioperative therapies in patients with high-risk muscle-invasive urothelial carcinoma and radical surgery will be collected.

Health-related quality of life (HRQoL) in patients with advanced renal cell carcinoma or advanced urothelial cancel will be evaluated for up to two years.

ELIGIBILITY:
Inclusion Criteria:

Cohorts aRCC and aUBC (prospective)

* Female and male patients with aRCC or aUBC (locally advanced, inoperable or metastatic)
* Patients at start of their first-line systemic treatment for aRCC or aUBC
* Written informed consent

  * Patients participating in the PRO module: signing of in-formed consent form and completion of baseline questionnaire before start of initial systemic treatment
  * Patients not participating in the PRO module: within twelve weeks after start of systemic first-line for aRCC or aUBC
* Age ≥ 18 years

Cohort High-risk MIUC (prospective and retrospective)

* Histologically proven muscle-invasive urothelial carcinoma (MIUC) of the lower or upper urinary tract (ICD-10 C65, C66, C67.x, C68.x). Mixed histologies are allowed (main compo-nent must be urothelial carcinoma, with minor variants accept-ed).
* Radical surgery (e.g., radical cystectomy, nephroureterecto-my) between October 1, 2021 and October 31, 2024.
* High-risk of recurrence, defined as follows: Post-operative, pathological tumor status

  * ypT2-ypT4 and/or ypN+ and without clinically detectable metastases (M0) at cystectomy for patients with prior neo-adjuvant chemotherapy or
  * pT3-pT4 and/or pN+ and without clinically detectable me-tastases (M0) at cystectomy for patients without prior neo-adjuvant chemotherapy.
* Age ≥ 18 years at the time of surgery.
* Written informed consent (only if patient is alive at time of data entry; not applicable for inclusion of deceased patients' data)

Exclusion Criteria:

Cohorts aRCC and aUBC (prospective)

* Patients with prior systemic therapy for aRCC or aUBC
* No systemic treatment for aRCC or aUBC

Cohort High-risk MIUC (prospective and retrospective)

* Partial cystectomy or partial nephrectomy of the primary tumor as definitive therapy
* Metastatic disease (M1) at the time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with locally advanced and inoperable, or metastatic Renal Cell Carcinoma (aRCC); locally advanced and inoperable, or metastatic Urothelial Cancer (including Bladder Cancer) (aUBC); or High-risk Muscle-Invasive Urothelial Carcinoma (High-risk MIUC)
Sampling Method: Non-Probability Sample
Enrollment: 1930 (Estimated)
Dates: Start 2017-12-07 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Course of treatment (treatment reality) | 3 years per patient
  Documentation of anamnestic data and therapy sequences

SECONDARY OUTCOMES:
Best Response | 3 years per patient
  Documentation of response rates per line of treatment.
Progression-free survival | 3 years per patient
  Documentation of progression-free survival per line of treatment.
Overall survival | 3 years per patient
  Documentation of overall survival time.
Health-related quality of life (Patient-reported outcome) | 2 years per patient
  Cohort aRCC: National Comprehensive Cancer Network/ Functional Assessment of Cancer Therapy (FACT)-Kidney Symptom Index 19 (NCCN-FACT FKSI-19) Cohort aUBC: NCCN/FACT Bladder Symptom Index (NCCN-FACT FBlSI-18, Version 2)
Treatment symptom related quality of life | 2 years per patient
  Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE™) - Items/Scores cohort aRCC: 3/7/15/22/24/27/28/50/51; Items/Scores cohort aUBC: 3/7/15/22/24/27/28/39/45/50/51

CONTACTS AND LOCATIONS:
Overall Officials: Michael Staehler, Prof. Dr., Study Chair — Ludwig Maximilian University of Munich, Dept. of Urology - University Hospital, Munich, Germany; Peter Goebell, Prof. Dr., Study Chair — University Clinic Erlangen, Department of Urology Comprehensive Cancer Center Erlangen EMN, Erlangen, Germany; Lothar Müller, Dr., Study Chair — Onkologie UnterEms, Leer-Emden-Papenburg, Leer, Germany; Viktor Grünwald, Prof. Dr., Study Chair — University Hospital Essen West German Cancer Center Essen, Clinic for Medical Oncology and Clinic for Urology, Essen, Germany; Carsten Grüllich, Prof. Dr., Study Chair — Sana Clinic Hof, Dept. of Hematology and Oncology, Hof, Germany; Christian Gratzke, Prof. Dr., Study Chair — University Hospital Freiburg, Dept. of Urology, Freiburg, Germany
Locations (1):
- Multiple sites, Germany, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No